CLINICAL TRIAL: NCT06820697
Title: Expanding Access to HIV Self-test Kits: Sustaining Private Sector Channels That Enable Access to Preventive Health Services
Brief Title: Private-sector Access to Testing for Health Sustainability
Acronym: PATHS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01MH136921 (NIH); R01MH136921 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HIV Prevention
Keywords: HIV; Tanzania; Pharmacies; AGYW; HIV self-test kits; adolescent girls and young women

STUDY DESIGN:
Intervention Model Description: Randomization of shops is at the ward level. Wards, and thus shops located in those wards, will be randomized to high or low HIVST kit subsidy groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High subsidy (Experimental): The high subsidy group will start off with a 90% subsidy for purchasing HIV self-test kits to sell in their shops.
  Interventions: Behavioral: High HIVST kit subsidy
- Low subsidy (Active Comparator): The low subsidy group will start off with a 50% subsidy for purchasing HIV self-test kits to sell in their shops.
  Interventions: Behavioral: Low HIVST kit subsidy

INTERVENTIONS:
Behavioral: Low HIVST kit subsidy — The two study groups are the "high" and "low" subsidy groups. The high subsidy group will start off with a 90% subsidy while the low subsidy group will start off with a 50% subsidy. Both study groups will experience decreasing subsidies at each phase of the study.
  Arms: Low subsidy
Behavioral: High HIVST kit subsidy — The two study groups are the "high" and "low" subsidy groups. The high subsidy group will start off with a 90% subsidy while the low subsidy group will start off with a 50% subsidy. Both study groups will experience decreasing subsidies at each phase of the study.
  Arms: High subsidy

SUMMARY:
New and innovative strategies are urgently needed to increase the uptake of HIV prevention and sexual and reproductive health services among adolescent girls and young women (AGYW) in sub-Saharan Africa. To ensure the real-world sustainability of free distribution of HIV self-test kits to AGYW by private drug shops and pharmacies, investigators will rigorously test supply-side subsidy structures for shopkeepers' provision of HIV-self test kits to AGYW combined with prosocial motivational supports. The combination of non-monetary and monetary support structures aims to emulate real-world health financing models for public-private partnerships and ultimately aims to improve equity in access to critical prevention services for AGYW at scale.

DETAILED DESCRIPTION:
This is an implementation-effectiveness trial that tests program adoption, implementation, and maintenance of free HIV self-test kit (HIVST) distribution to adolescent girls and young women (AGYW) financed by profits from HIVST kit sales to non-AGYW customers. To initiate adoption, the study will offer pharmacy and drug shopkeepers the opportunity to procure subsidized HIVST to simultaneously distribute to AGYW for free (reimbursed by the study mimicking government-supported provision) and sell to non-AGYW customers for profit, gradually phasing out procurement subsidies over 36 months to test maintenance of the segmented pricing model for real-world sustainability (Aim 1). Investigators will implement non-monetary motivation boosters to sustain shopkeeper engagement over the study period and use mixed-methods to understand shopkeepers' experiences and necessary conditions for program maintenance and provider behavior change (Aim 2), which will inform the co-design of a progressive scale-up plan to achieve national coverage with Tanzanian AGYW, public, and private partnership stakeholders (Aim 3). At the study's conclusion, investigators will have a comprehensive understanding of the support structures shops need to sustain HIVST kit provision for AGYW. Importantly, the study will contribute to generalizable learning about the structures required for commercially sustainable public-private partnerships for high-impact public health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Owners/staff of retail drug shops and pharmacies located in the study regions
* Age 18 and older

Exclusion Criteria:

* Refusal to install and track sales and distribution of HIVST kits using the Maisha Meds data system provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of HIVST kits distributed to AGYW per shop month | 39 months
  HIVST kit distribution per shop per month will be tracked via Maisha Meds sales and inventory management system. The data from Maisha Meds will include a tag that identifies the kit recipient as an AGYW and will include the price paid for the HIVST kit ($0 for AGYW).

SECONDARY OUTCOMES:
Adoption | 39 months
  Proportion of shops continuing to procure HIVST kits throughout the study
Implementation 1 | 39 months
  Proportion of shops that offer free HIVST to AGYW mystery client actors
Implementation 2 | 39 months
  Proportion of shops continuing to provide free HIVST throughout the study period
Implementation 3 | 39 months
  Shopkeeper perspectives on challenges and successes related to providing HIVST kits free to AGYW as measured via surveys and in-depth interviews.
Maintenance | 39 months
  Proportion of shopkeepers who intend to continue to purchase and sell HIVST kits; Shopkeeper and stakeholder perspectives on subsidies, reimbursements, and sustainability; Reasons for discontinuing the sale of HIVST kits; Proportion of shops continuing to purchase and sell HIVST kits after subsidies end
Implementation 4 | 39 months
  Proportion of shops that sell HIVST to non-AGYW mystery client actors

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Liu, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Mwanza Intervention Trials Unit, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
This project will produce survey data, in-depth interview transcripts, and product sales and distribution data. All data will be de-identified prior to receipt by the repository, but the information needed to generate a global unique identifier (GUID) for the NIMH Data Archive (NDA) will be collected for each subject if possible. This information includes First Name, Middle Name, Last Name, Sex, Date of Birth, City/Municipality of Birth. Because investigators are collecting data from participants in Tanzania, some of this information may be unavailable or may not meet the requirements for the GUID. In that case, pseudoGUIDs will be utilized.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The research community will have access to data when the award ends. As required by NDA, studies will also be created that contain the data used for every publication. Those studies will be shared when the pre-print is available. NDA studies have digital object identifiers (DOI) to aid in findability. Investigators will include that DOI in relevant publications. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.
Access Criteria: To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.